CLINICAL TRIAL: NCT04215575
Title: Baerveldt Glaucoma Implant Versus Ahmed Glaucoma Implant in One- Year Follow up, Comparative Study
Brief Title: Baerveldt (BGI) Valve Versus Ahmed(AGV) Valve in Management of Difficult Glaucoma Cases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, khaled hamdi elbaklish, principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FWA000017585 FMASU21/2017
Record Dates: First submitted 2019-12-29; First posted 2020-01-02 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Glaucoma, Open-Angle; Glaucoma Secondary; Glaucoma, Neovascular; Glaucoma, Angle-Closure
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma, Neovascular; Glaucoma, Angle-Closure

STUDY DESIGN:
Intervention Model Description: Participants were randomized to BGI model 101-350 placement (BGI group) or an AGV model FP7or S2 placement (AGV group). Follow-up visits were scheduled 1 day, 1 week, 1 month, 3 months, 6 months, 1 year postoperatively. The primary outcome measure was failure that defined as IOP >16 mmHg or less than a 20% reduction below baseline on 2 consecutive study visits.The IOP, the use of glaucoma medications, visual acuity (VA), visual fields, bleb morphology and rates of surgical complications were secondary outcome measures.
Who Masked: Participant, Investigator
Masking Description: A clinical trial design strategy in which parties involved in the trial, the investigator and participants, do not know which participants have been assigned which interventions. Type of masking include: double-blind masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BGI model 101-350 placement (BGI group) (Active Comparator): A 350 mm2 Baerveldt glaucoma implant was placed. Follow-up visits were scheduled 1 day, 1 week, 1 month, 3 months, 6 months, 1 year postoperatively. The primary outcome measure was failure that defined as IOP >16 mmHg or less than a 20% reduction below baseline on 2 consecutive study visits.The IOP, the use of glaucoma medications, visual acuity (VA), visual fields, bleb morphology and rates of surgical complications were secondary outcome measures.
  Interventions: Device: glaucoma implant procedure (Baerveldt)
- AGV model FP7 or S2 placement (AGV group) (Experimental): A 184 mm2 Ahmed glaucoma implant was placed. Follow-up visits were scheduled 1 day, 1 week, 1 month, 3 months, 6 months, 1 year postoperatively. The primary outcome measure was failure that defined as IOP >16 mmHg or less than a 20% reduction below baseline on 2 consecutive study visits. The IOP, the use of glaucoma medications, visual acuity (VA), visual fields, bleb morphology and rates of surgical complications were secondary outcome measures
  Interventions: Device: glaucoma implant procedure (Ahmed)

INTERVENTIONS:
Device: glaucoma implant procedure (Baerveldt) — A 350 mm2 Baerveldt glaucoma implant was placed in the superotemporal quadrant in 25 patients randomized to BGI group. A limbus-based conjunctival flap was dissected, and the implant was sutured to sclera 10 mm posterior to the limbus. A scleral graft was used to cover the limbal portion of the tube, and the conjunctiva was closed.
  Other Names: glaucoma valve surgery
  Arms: BGI model 101-350 placement (BGI group)
Device: glaucoma implant procedure (Ahmed) — A 184 mm2 Ahmed glaucoma implant was placed in the superotemporal quadrant in 56 patients randomized to AGV group. A fornix-based conjunctival flap was dissected, and the implant was sutured to sclera 10 mm posterior to the limbus. The Ahmed tube left patent and viscoelastic substance injected into anterior chamber. A scleral graft was used to cover the limbal portion of the tube, and the conjunctiva was closed.
  Other Names: glaucoma valve surgery
  Arms: AGV model FP7 or S2 placement (AGV group)

SUMMARY:
Refractory glaucoma is a difficult subject as many glaucoma devices attempt to reduce IOP. Baerveldt implant is considered as a large implant, and, on the contrary, Ahmed implant is considered a small implant as many comparisons have showed. Investigators have previously used two models S2 and FP7 Ahmed implant. Currently, investigators use Baerveldt implant in refractory glaucoma cases in order to compare it with the Ahmed implant.

DETAILED DESCRIPTION:
Eighty-one participants with glaucoma after ocular surgery or secondary glaucoma with persistent and uncontrolled IOP > 21 mmHg were randomized for placement of Baerveldt implant or Ahmed implant models using a standardized surgical technique.

The primary outcome was failure, which was defined as IOP >16 mmHg with glaucoma medication on 2 consecutive study visits. Secondary outcomes were IOP, medication use, visual acuity, complications, and interventions.

ELIGIBILITY:
Inclusion Criteria:

1 - patients with glaucoma who underwent a previous failed trabeculectomy or other intraocular surgery.

2- patients who had secondary glaucoma and are known to have a high failure rate with trabeculectomy such as neovascular, uveitis, or iridocorneal endothelial syndrome-associated glaucoma, were included in the study.

Exclusion Criteria:

1 - patients lacked light perception, unwilling or unable to give informed consent, were expected to be unavailable for follow-up visits.

2-had previous aqueous shunt implanted in the same eye, other external impediment to supero-temporal drainage device implantation.

3- presence of silicone oil, vitreous in the anterior chamber sufficient to require a vitrectomy.

4-uveitis associated with a systemic condition like juvenile rheumatoid arthritis, nanophthalmos, Sturge-Weber syndrome or other conditions associated with elevated episcleral venous pressure.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-20 (Actual)

PRIMARY OUTCOMES:
IOP | one year follow up
  mean IOPs
glaucoma medications | one year follow up
  mean number of glaucoma medications

SECONDARY OUTCOMES:
visual acuity | one year follow up
  log MAR Snellen median and interquartile Range values

IPD SHARING:
Plan to Share IPD: No
no actual plan

REFERENCES:
- [Derived] Elbaklish KH, Saleh SM, Gomaa WA. Baerveldt Glaucoma Implant versus Ahmed Glaucoma Implant in a One-Year Follow Up, Comparative Study. Clin Ophthalmol. 2020 Jan 8;14:29-39. doi: 10.2147/OPTH.S224654. eCollection 2020. PMID 32021066